CLINICAL TRIAL: NCT00301366
Title: Multi-center, Open-label Trial to Evaluate the Safety and Tolerability of Alpha-1 MP in Subjects With Alpha-1-antitrypsin (AAT) Deficiency
Brief Title: The Safety and Tolerability of Alpha-1 Modified Process (MP) In Subjects With Alpha-1-antitrypsin (AAT) Deficiency
Acronym: STAMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11815
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: alpha 1-Antitrypsin Deficiency; alpha 1-Antitrypsin; pulmonary emphysema
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Emphysema | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alpha-1 Proteinase Inhibitor (Human), modified process (Experimental): Study the safety and tolerability of weekly infusions of Alpha-1 Proteinase Inhibitor (Human), modified process (Alpha-1 MP, 60 mg/kg) over 20 weeks of therapy in adult Alpha-1 antitrypsin deficient subjects.
  Interventions: Drug: alpha-1 proteinase inhibitor (human)

INTERVENTIONS:
Drug: alpha-1 proteinase inhibitor (human) — 60 mg/kg weekly for 20 weeks
  Other Names: Prolastin; Alpha-1 antitrypsin (AAT); BAY x 5747; BAY 10-5233; TAL-05-00007

SUMMARY:
The purpose of this clinical study is to assess the safety and tolerability of Alpha-1 MP in adult Alpha1-antitrypsin deficient patients.

DETAILED DESCRIPTION:
The objective of this clinical trial (STAMP: Safety and Tolerability of Alpha-1 Modified Process) is to study the safety and tolerability of Alpha-1 MP in adult Alpha 1-antitrypsin deficient subjects as reported over 20 weeks of therapy. The primary objective is to describe the nature and frequency of treatment-emergent adverse events with "treatment-emergent" defined as any adverse event occurring after the start of the first study drug infusion.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of congenital Alpha1-antitrypsin deficiency
* Documented forced expiratory volume in 1 second (FEV1 ) between 20% - 80% of predicted value within last 6 months.
* Signed written informed consent prior to initiation of any study related procedures.

Exclusion Criteria:

* Females who are pregnant, breast feeding, or if of child-bearing potential, unwilling to practice adequate contraception throughout the study
* Use of systemic steroids within the 2 weeks prior to receiving study treatment (this does not include the use of inhaled steroids used on a routine or as needed basis).
* Subjects who have had exacerbations of their disease within one month of trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hanna, MSc, Study Director — Grifols Therapeutics LLC
Locations (10):
- United States (8):
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - St Lukes-Roosevelt Hospital Center, New York, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Center at Tyler, Tyler, Texas
- United Kingdom (2):
  - University of Cambridge - Cambridge Institute for Medical Research, Cambridge, England
  - University Teaching Hospital of Edinburgh, Edinburgh, Scotland

REFERENCES:
- [Background] Wewers MD, Casolaro MA, Sellers SE, Swayze SC, McPhaul KM, Wittes JT, Crystal RG. Replacement therapy for alpha 1-antitrypsin deficiency associated with emphysema. N Engl J Med. 1987 Apr 23;316(17):1055-62. doi: 10.1056/NEJM198704233161704. PMID 3494198
- [Background] Gadek JE, Klein HG, Holland PV, Crystal RG. Replacement therapy of alpha 1-antitrypsin deficiency. Reversal of protease-antiprotease imbalance within the alveolar structures of PiZ subjects. J Clin Invest. 1981 Nov;68(5):1158-65. doi: 10.1172/jci110360. PMID 7028785
- [Background] Gadek JE, Fells GA, Zimmerman RL, Rennard SI, Crystal RG. Antielastases of the human alveolar structures. Implications for the protease-antiprotease theory of emphysema. J Clin Invest. 1981 Oct;68(4):889-98. doi: 10.1172/jci110344. PMID 6169740
- See also: The "Alpha-1 Foundation", dedicated to providing the leadership and resources that will result in increased research, improved health, worldwide detection and a cure for Alpha-1 Antitrypsin Deficiency — http://www.alphaone.org
- See also: AlphaNet, Inc devoted to improving the lives of individuals with Alpha-1 antitrypsin deficiency through comprehensive disease management services, clinical research administration, and consultative services — http://www.alphanet.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First-subject-first-dose was 12 June 2006, last-subject-last-visit was 20 March 2007. The study was performed in 10 clinical sites, 8 sites in the United States and 2 sites in the United Kingdom.
Groups:
- Alpha-1MP Treatment Group: All subjects received open-label weekly IV infusions of 60 mg/kg body weight of functional Alpha-1 MP for 20 weeks
Period: Overall Study
Arm/Group | Alpha-1MP Treatment Group
Started | 38
Completed | 37
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entered Study
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 35
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs) Defined as Any Adverse Event (AE) Occurring During or After the Start of the First Study Drug Infusion.
Description: An adverse event is any untoward medical occurrence in a subject or clinical investigation subject administered with a pharmaceutical product. The adverse event does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the medicinal product.
Time Frame: 24 weeks
Population: 38 subjects received study medication and one subject discontinued from the study due to an AE. Therefore, 37 subjects completed the study. 18 subjects were naive ((i.e., never having received previous Alpha-1 protease inhibitor augmentation therapy) and 19 subjects were non-naive.
Measure: Number; unit: Participants
Arm/Group | Alpha-1 MP Treatment Group
Number analyzed (Participants) | 38
Participants
  Number of Participants Analyzed | 38
  Subjects experiencing TEAEs | 26
  Subjects with TEAEs <24 hrs. of A-1 MP infusion | 17
  Alpha-1 MP subjects with ≥1 drug-related TEAE | 5

ADVERSE EVENTS:
Arm/Group | Alpha-1MP Treatment Group
Serious Adverse Events (participants affected / at risk) | 2/38
Other Adverse Events (participants affected / at risk) | 26/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1MP Treatment Group (N=38)
Pneumonia (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1MP Treatment Group (N=38)
Nausea (Gastrointestinal disorders) | 6 (6)
Chest pain (General disorders) | 4 (4)
Influenza like illness (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot flush (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor, thirty days in advance of submission, in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution that satisfies both parties.